CLINICAL TRIAL: NCT06678230
Title: Multicenter, Single-Arm, Phase II Clinical Trial of Eribulin in Combination with Anrotinib for HER-2 Negative Locally Advanced or Metastatic Breast Cancer.
Brief Title: Clinical Trial of Eribulin in Combination with Anrotinib for HER-2 Negative Locally Advanced or Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-HS-061
Record Dates: First submitted 2024-01-01; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: Eribulin; Anlotinib
MeSH Terms: conditions — Breast Neoplasms | interventions — anlotinib; eribulin

STUDY DESIGN:
Intervention Model Description: Alibulin 1.4mg/m2, D1, 8; Every 3 weeks is a cycle; Androtinib 12mg, QD, po, applied for 14 days, stopped for 7 days, and every 3 weeks was a cycle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- This is a single-arm, single-center, phase II clinical trial of eribulin in combination with erlotin (Experimental): This trial is planned to enroll 40 subjects with HER-2 negative locally advanced or metastatic breast cancer who have received prior chemotherapy with anthracyclines and paclitaxel, treated with eribulin in combination with erlotinib.
  Trial drug: eribulin 1.4 mg/m2, D1,8; one cycle every 3 weeks; Amlotinib 12 mg, QD, po, applied for 14 days and stopped for 7 days, one cycle every 3 weeks.
  All subjects will receive long-term dosing until intolerable toxicity or disease progression or death or voluntary withdrawal or the end of this trial (meaning completion of the trial or early termination of the trial).
  During the treatment period, all subjects will be evaluated for antitumor efficacy every 6 weeks and disease status will be determined by the investigator according to RECIST 1.1 criteria until disease progression or death or refusal to come to the hospital for follow-up or the end of the trial (meaning completion of the trial or early termination of the trial), whichever event occurs
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — Alibulin 1.4mg/m2, D1, 8; Every 3 weeks is a cycle; Androtinib 12mg, QD, po, applied for 14 days, stopped for 7 days, and every 3 weeks was a cycle.
  Other Names: Eribulin

SUMMARY:
Study Objective: To evaluate the progression-free survival of HER-2 negative locally advanced or metastatic breast cancer subjects treated with eribulin in combination with erlotinib Trial Drug: Erlotinib Targets: Erlotinib is a novel small-molecule multi-targeted tyrosine kinase inhibitor, which can inhibit the kinase activities of vascular endothelial growth factor receptor (VEGFR1-3), platelet-derived growth factor receptor (PDGFRα, PDGFRβ), fibroblast growth factor receptor (FGFR1-4), stem cell growth factor receptor, etc., and thus exert anti-tumor angiogenesis, thereby exerting anti-tumor angiogenesis and anti-vascularity. PDGFRα, PDGFRβ), fibroblast growth factor receptor (FGFR1-4), stem cell growth factor receptor and other kinase activities, and then play the role of anti-tumor angiogenesis and inhibition of tumor growth. Results of previous studies, known efficacy and adverse effects: The single-agent regimen of amlotinib has been clinically approved in non-small cell lung cancer, gastric cancer, and soft tissue sarcoma. In breast cancer, the II clinical study of amlotinib monotherapy for the treatment of HER-2 negative advanced breast cancer in the second line and above showed that the PFS of amlotinib monotherapy was 5.22 months, ORR was 15.4%, and DCR was 80.8%, which demonstrated that amlotinib has better anti-tumor activity. Major adverse reactions: fatigue, weight loss, hypertension, diarrhea, nausea, vomiting, hematemesis

DETAILED DESCRIPTION:
This is a single-arm, single-center, Phase II clinical trial of eribulin in combination with amlotinib in subjects with HER-2 negative locally advanced or metastatic breast cancer.

The trial is planned to enroll 40 subjects with HER-2 negative locally advanced or metastatic breast cancer who have received prior chemotherapy with anthracycline and paclitaxel-based agents to receive eribulin in combination with erlotinib.

Trial drug: eribulin 1.4 mg/m2, D1,8; one cycle every 3 weeks; Amlotinib 12 mg, QD, po, applied for 14 days and stopped for 7 days, one cycle every 3 weeks.

All subjects will receive long-term dosing until intolerable toxicity or disease progression or death or voluntary withdrawal or the end of this trial (meaning completion of the trial or early termination of the trial).

During the treatment period, all subjects will be evaluated for antitumor efficacy every 6 weeks and disease status will be determined by the investigator according to RECIST 1.1 criteria until disease progression or death or refusal to come to the hospital for follow-up or the end of the trial (meaning completion of the trial or early termination of the trial), whichever event occurs first. After a subject's disease progression or refusal to come to the hospital for follow-up, the investigator will make a telephone visit every 3 months (each month will be counted as 30 days) to obtain information about the subject's survival, whether he/she is receiving other antitumor therapy, etc.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed breast cancer.
* immunohistochemistry HER-2 negative at this center
* subjects with locally recurrent or metastatic breast cancer who have received chemotherapy with anthracyclines and paclitaxel prior to the current chemotherapy regimen. Treatment prior to study entry must meet the following criteria: a. The regimen must include anthracyclines (e.g., doxorubicin, epirubicin, piroxicam) and paclitaxel (e.g., paclitaxel, docetaxel) in any combination or other order of administration. If these drugs are contraindicated in the intended subject, prior use of these drugs in prior therapy is not required but is documented in the subject's medical history. b. Some of these regimens may be used as adjuvant and/or neoadjuvant therapies, and subjects may also have been previously treated with anti-estrogenic agents. c. ≤2 lines of chemotherapy targeting recurrent/metastatic lesions: i Anthracyclines and paclitaxel adjuvant therapy within 12 months of progression; ii progression on advanced first/second line therapy; iii subjects must have demonstrated disease progression on the most recent chemotherapy.
* Endocrine therapy targeting recurrent/metastatic lesions will not be counted towards the number of lines of therapy.
* Measurable lesions meet the following criteria:Exclusion Criteria:a. At least one lesion with a longest diameter ≥1.0 cm for non-lymph nodes or a short-axis diameter ≥1.5 cm for lymph nodes, which can be measured serially using computed tomography/magnetic resonance imaging (CT/MRI) according to RECIST 1.1. b. If only one target lesion is non-lymph node, its longest diameter should be ≥1.5 cm. Physical Status Score ≤ 2.
* Age ≥ 18 and ≤ 70 years at the time of signing the informed consent form.
* Appropriate renal function as evidenced by serum creatinine ≤ 2.0 mg/dL, or serum creatinine clearance ≥ 40 mL/min according to the Cockcroft-Gault formula.
* Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L, hemoglobin ≥ 9.0 g/dL, and platelet count ≥ 100 x 109/L as evidence of adequate bone marrow function.
* Bilirubin ≤ 1.5 times the upper limit of normal (ULN); and alkaline phosphatase (ALP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤ 3.0 times the ULN (≤ 5.0 times the ULN in the case of hepatic metastases) as evidence of adequate bone marrow function. 5.0 times upper limit of normal) as evidence of appropriate liver function.
* Subjects are willing and able to comply with the study protocol throughout the study period.
* All female subjects will be considered of childbearing potential unless postmenopausal (at least 12 consecutive months of amenorrhea, in the appropriate age group, and with no other known or suspected cause) or surgically sterilized (i.e., ≥1 menstrual cycle of bilateral tubal ligation, or hysterectomy and/or bilateral oophorectomy prior to randomization). Female subjects of childbearing potential must agree to use two highly effective methods of contraception beginning with their last menstrual period prior to randomization grouping (or until two highly effective methods of contraception have been used for at least one menstrual cycle using the double-barrier method described below), during the study period, and for a period of 3 months after the final dose of study treatment. Female subjects exempted from this requirement were subjects who were completely abstinent. If currently abstinent, the subject must agree to use a double barrier method of contraception (i.e., condom with spermicide and an occlusive cap (uterine cap or cervical/vault cap)) if she becomes sexually active during the study treatment period, or two highly effective methods of contraception for at least one menstrual cycle and until 3 months after the final dose of study treatment. Highly effective methods of contraception include: a. Implantable intrauterine device (IUD) or contraceptive system, b. Barrier methods of contraception: spermicide-containing condom or occlusive cap (uterine cap or cervix/fornix cap), and c. Recognized hormonal contraceptive methods: oral, injectable, or implantable. Female subjects using hormonal contraceptives must receive a stable dose of the same hormonal contraceptive product from the last menstrual period prior to randomization and must continue to use the same hormonal contraceptive product for the duration of the study treatment as well as for 3 months after the final dose of study treatment, d. Confirmed azoospermic vasectomy partner.
* Voluntarily agrees to, and signs, a written informed consent form, and is willing and able to comply with all aspects of the trial protocol, and the patient may withdraw consent at any time without prejudice.

Exclusion criteria：

* previous neoadjuvant or adjuvant therapy containing eribulin (anitrotinib may have been applied)
* patients in whom anitrotinib is contraindicated.
* patients with active symptomatic brain metastases or meningeal metastases.
* patients with active/refractory infections requiring ongoing anti-infective therapy.
* pulmonary lymphovascular dissemination resulting in pulmonary dysfunction requiring active therapy, including the use of oxygen.
* severe cardiovascular impairment (history of congestive heart failure greater than New York Heart Association (NYHA) class II), unstable angina pectoris or myocardial infarction within the past 6 months, or severe cardiac arrhythmias.
* Subjects with allogeneic organ transplants requiring immunosuppressive therapy.
* Subjects known to be positive for Human Immunodeficiency Virus (HIV).
* Subjects with prior malignant tumors other than breast, cervical carcinoma in situ, and non-melanoma skin cancer. Subjects with a prior malignancy other than breast cancer and non-melanoma skin cancer, unless the prior malignancy has been previously diagnosed and definitively treated for at least 5 years without evidence of subsequent recurrence.
* Subjects with pre-existing neuropathy > Grade 2.
* Subjects with hypersensitivity to chondroitin B and/or chemical derivatives of chondroitin B.
* Any medical condition that, in the opinion of the Investigator, makes a subject ineligible for entry into the study.
* Subjects with a known human immunodeficiency virus (HIV)-positive condition.
* Subjects with a known human immunodeficiency virus (HIV)-positive condition.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 33 months
  PFS, commonly referred to in medicine as progression-free survival, is the main indicator used to measure the effectiveness of agents used to treat a tumour during the course of treatment, and is commonly used to assess the treatment of cancer patients, with a strong correlation to overall survival, usually measured in months.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center, The First Affiliated Hospital of Jilin University, Changchun, Jilin Province, China, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided